CLINICAL TRIAL: NCT00002543
Title: GALLIUM NITRATE FOR THE TREATMENT OF MALIGNANT TUMORS, A PHASE I STUDY
Brief Title: Gallium Nitrate in Treating Children With Brain Tumor, Neuroblastoma, Rhabdomyosarcoma, Non-Hodgkin's Lymphoma, or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MCW-ARRC-22393; CDR0000063244 (Registry Identifier: PDQ (Physician Data Query)); CHW-93/59; NCI-T93-0097D
Record Dates: First submitted 1999-11-01; First posted 2004-10-05 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2007-05

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma; Neuroblastoma; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: recurrent childhood rhabdomyosarcoma; recurrent childhood brain tumor; recurrent neuroblastoma; recurrent childhood lymphoblastic lymphoma; unspecified childhood solid tumor, protocol specific; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Neuroblastoma; Sarcoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — gallium nitrate

INTERVENTIONS:
Drug: gallium nitrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: : Phase I trial to study the effectiveness of gallium nitrate in young patients who have malignant brain tumors, neuroblastoma, rhabdomyosarcoma, non-Hodgkin's lymphoma, or refractory solid tumor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and side effects of gallium nitrate (GAN) when used as an anticancer agent in pediatric patients with refractory solid tumors, including malignant brain tumors, neuroblastoma, rhabdomyosarcoma, and non-Hodgkin's lymphoma. II. Evaluate these side effects in these patients.

OUTLINE: Single-Agent Chemotherapy. Gallium Nitrate, GAN, NSC-15200.

PROJECTED ACCRUAL: At least 3 patients will be accrued at each dose studied.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven rhabdomyosarcoma, non-Hodgkin's lymphoma, or other solid tumor refractory to conventional therapy or for which no effective curative therapy is known Re-biopsy required if disease recurs more than 2 years after initial diagnosis recommended if radiographic abnormalities suggest tumor recurrence within 5 months of completing radiotherapy or chemotherapy

PATIENT CHARACTERISTICS: Age: 21 and under at diagnosis Performance status: Karnofsky 50%-100% Life expectancy: More than 4 weeks Hematopoietic: (unless extensive bone marrow involvement) ANC greater than 750 Platelets greater than 75,000 Hepatic: Not specified Renal: Creatinine normal for age OR Glomerular filtration rate at least 50 mL/min per 1.73 square meters Other: Adequate nutritional status No serious uncontrolled infection No pregnant or nursing women

PRIOR CONCURRENT THERAPY: At least 2 weeks since other anticancer therapy and recovered Prior radiotherapy or surgery for symptomatic lesions allowed provided site of evaluable disease remains untreated Prior bone marrow or stem cell transplantation allowed No concurrent anticancer therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Estimated)
Dates: Start 1995-02; Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry T. Whelan, MD, Study Chair — Medical College of Wisconsin
Locations (3):
- United States (3):
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Medical College of Wisconsin, Milwaukee, Wisconsin